CLINICAL TRIAL: NCT00058799
Title: Treatment of High Risk Acute Leukemia With CD40 Ligand and IL-2 Gene Modified Autologous Skin Fibroblasts and Tumor Cells
Brief Title: Treating High Risk Leukemia With CD40 Ligand & IL-2 Gene Modified Tumor Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Dist Serv Prof, Center for Gene Therapy, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H6408-Leu Leu
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): Patients are treated with up to six injections of their gene-modified CD40L and IL-2 skin fibroblasts and leukemic blasts, separated by one-two weeks in an immunological treatment window.
  Interventions: Biological: Dose Level 1
- Dose Level 2 (Experimental): Patients are treated with up to six injections of their gene-modified CD40L and IL-2 skin fibroblasts and leukemic blasts, separated by one-two weeks in an immunological treatment window.
  Interventions: Biological: Dose Level 2
- Dose Level 3 (Experimental): Patients are treated with up to six injections of their gene-modified CD40L and IL-2 skin fibroblasts and leukemic blasts, separated by one-two weeks in an immunological treatment window.
  Interventions: Biological: Dose Level 3

INTERVENTIONS:
Biological: Dose Level 1 — Leukemic Blasts 2 x 10^7; IL-2 Fibroblasts 2 x 10^7; CD40L Fibroblasts 2 x 10^5
  Arms: Dose Level 1
Biological: Dose Level 2 — Leukemic Blasts 2 x 10^7; IL-2 Fibroblasts 2 x 10^7; CD40L Fibroblasts 2 x 10^5
  Arms: Dose Level 2
Biological: Dose Level 3 — Leukemic Blasts 2 x 10^7; IL-2 Fibroblasts 2 x 10^7; CD40L Fibroblasts 4.2 x 10^7
  Arms: Dose Level 3

SUMMARY:
This research study is to determine the safety and dosage of special cells that may make the patients own immune system fight the leukemia. To do this we will put special genes into cells called fibroblasts that we have grown in the laboratory from a skin sample. The genes we put in these fibroblasts make them produce substances called CD40 Ligand (CD40L) and interleukin-2 (IL-2). These are natural substances that may help the immune system kill leukemia cells. Some of these fibroblasts producing CD40L and IL-2 mixed with a small quantity of the leukemic cells will then be put back into the body.

Studies of cancers in animals and in cell lines suggest that substances like CD40L and IL-2 when mixed with cancer cells do help the body to recognize and kill these cancer cells. A treatment using IL-2 has been previously used in more than 40 children with neuroblastoma and similar treatments are being used in adults with other cancers. Some of the patients have shown significant tumor responses. However, we do not know if this treatment will work and we do not know the right amount of each of the special cells to use, so different patients will get different combination and numbers of cells.

The purpose of this study is to learn the side effects and safe dosage of these special cells.

DETAILED DESCRIPTION:
Before starting in the treatment part of this study, leukemia cells and skin fibroblasts will be collected from the patient - called "procurement" - to allow us to make the vaccine. These leukemia cells are taken from either peripheral blood, leukopheresis product or bone marrow. The fibroblasts will be prepared in the laboratory with specially produced human viruses (adenoviruses) that carry the IL-2 or the CD40L gene. The viruses will "drop off" the genes inside the fibroblasts. The CD40L and IL-2 genes are meant to help stimulate the immune system to fight the leukemia. The modified fibroblasts will be injected with a number of leukemic cells under the skin. All the cells will be irradiated before injection to stop them growing. Patients will receive three shots. Depending on the response, patients may be able to have three additional shots.

In order to collect the skin fibroblasts at the very beginning of the study, and then during the study, we will perform small skin biopsies. In particular before the second shot, and then again about 1 week later, we will look for both the modified and leukemia cells that have been re-injected under the skin. We will do this by taking a skin biopsy from the place where the cells were injected. The area where the skin biopsy will be obtained will be sterilized and then numbed with a local acting agent. The skin will be removed with a "tissue punch" which will cut a circle of approximately 1/4th of an inch into the skin. The site where the skin was removed will be closed with suture, tape or stitches. The area will be covered with dry gauze and adhesive tape. These tests are to see whether the shots are killing leukemia cells and to make sure leukemia cells are not growing at the injection site.

To study how the immunity is working in the system, we will take blood samples before first injection, then weekly for 10 weeks, on week 12, once a month for a year, and then eventually once a year for fifteen years. These samples will be approximately 1 tablespoons of blood, which is considered a safe amount. If the patient has additional injections, blood will be drawn prior to each injection. Additional office visits may be necessary.

Also, patients will need to have a bone marrow test before enrolling on the study and at week 12. If the patient is not responding, they may have treatment with other chemotherapy or radiation. Patients will need to come to the clinic on the days of blood drawing and to be seen at Texas Children's Cancer Center/The Methodist Hospital at weekly intervals for 10 weeks, then every other week for 6 weeks, and then monthly for a year. Thereafter, patients will either be seen in the clinic or contacted by one of the research staff working on this study once a year for 15 years. Additional visits may be necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Patients less than or equal to 75 years old with lymphoid (pre-B, B, T, non B-, non T, or Burkitt if bone marrow blasts > 20%) or acute myeloid leukemia (M0 to M7) or myelodysplastic syndrome and with: Disease that has entered remission with chemotherapy and/or bone marrow transplantation, but is considered to be at high risk of relapse. or Primary, or relapsed treatment-refractory disease who, at the time of reinjection of the tumor vaccine, are at a state of complete or partial cytological remission disease (<20% blasts infiltrating the bone marrow) after a second/higher line of conventional and/or high dose chemotherapy.
2. Patients must have a life expectancy of at least 10 weeks.
3. Patients must have ECOG performance status of 0-2 as below:
4. Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study, and have an absolute neutrophil count >500/mm3, absolute lymphocyte count >200/mm3, and platelet count >50,000/mm3.
5. Patients must not have active GvHD at the time of protocol entry.
6. Patient has not received high dose steroids within the last week or other immunosuppressive drugs within a week (or longer as indicated by the half life of the agent)
7. Patients must not be infected at time of protocol entry, and should not be receiving antibiotics (other than prophylactic Septra.)
8. Patients must not be HIV-positive.
9. Patients must have adequate liver function (bilirubin<1.5 mg% SGOT<2x normal, normal prothrombin time).
10. Patients must have transduced cells available that are demonstrably >20% CD40L expressing fibroblasts and producing>150 pg IL-2/10 6 cell/24 hr.
11. Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.
12. Patient must not have received treatment with other investigational agents within the last 4 weeks.
13. Patients must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom.

Exclusion Criteria:

1. Rapidly progressive/refractory disease (>20% blasts infiltrating the bone marrow)
2. Life expectancy < 10 weeks
3. Active infection
4. Need for concomitant drugs except analgesics
5. Pregnancy or lactation
6. Seropositive for HIV

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1999-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
• To determine the safety of up to six subcutaneous (SC) injections of autologous tumor cells admixed with autologous gene-modified skin fibroblasts. These fibroblasts are modified ex vivo to express the human CD40 Ligand (hCD40L) and interleukin-2 (hIL | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Texas Children's Hospital GCRC, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas